CLINICAL TRIAL: NCT00792220
Title: "Mobile Stroke-Unit" for Reduction of the Response Time in Ischemic Stroke
Acronym: MSU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Saarland (Other)
Collaborators: Deutsches Rotes Kreuz DRK-Blutspendedienst Baden-Wurttemberg-Hessen (Other); Meytec Information Systems GmbH, Werneuchen (Unknown); Else Kröner Fresenius Foundation (Other); Mercedes-Benz AG, Niederlassung Saarbrücken (Unknown); Stadt Homburg (Unknown); Rettungsstiftung Saarland (Unknown); Rettungsdienst Logistik-Service GmbH, Saarland (Unknown)
Responsible Party: Prof. Dr. med. Klaus Fassbender, University Hospital of the Saarland, Department of Neurology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSU
Record Dates: First submitted 2008-11-13; First posted 2008-11-17 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Stroke
Keywords: stroke; mobile stroke unit; thrombolysis; stroke management; computerized tomography
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MSU (Experimental)
  Interventions: Procedure: MSU
- OCCM (Active Comparator)
  Interventions: Procedure: OCCM

INTERVENTIONS:
Procedure: MSU — In the "Mobile Stroke Unit" procedure: Conventional Emergency Medical Service together with the MSU will meet at the side, where the patient is found. The MSU is an ambulance, equipped with a neurologist and neuroradiologist and includes CT scanner and point of care laboratory unit. The patient's medical history and the physical examination will be directly performed by the neurologist. CT scan analysis will be performed by the neuroradiologist, while the neurologist will analyze the blood samples with the point of care laboratory unit. If the inclusion and exclusion criteria are fulfilled, the thrombolytic therapy will directly be started by the neurologist. A possible thrombolytic therapy will be performed under the current inclusion and exclusion criteria that are associated with the rt-PA drug approval in Europe. After performance of the acute therapy, the patient will be transported to the University Hospital of the Saarland.
  Arms: MSU
Procedure: OCCM — In the optimized conventional clinical management: After patient's medical history, physical examination and emergency treatment by the emergency physician, the patient will be transported to the University Hospital of the Saarland. The delivery of the patient will directly take place at the CT scanner. The neurologist will perform a second medical history, physical examination, while the blood will be drawn by the assisting nurse. CT scan will be performed, while the blood will be analyzed by point of care technique, placed close to the CT scanner. Additionally the blood will be sent in parallel to the hospital central laboratory for conventional laboratory analysis. Depending on the results, a thrombolytic therapy will be initiated directly at the CT. Thereafter, the patient will be transported to the hospital Stroke Unit.
  Arms: OCCM

SUMMARY:
Stroke, the most common cause of permanent disability, the second most common cause of dementia and third most common cause of death, has tremendous socio-economic consequences.

Currently, systemic thrombolysis with the tissue plasminogen activator represents the only causal and approved treatment for acute ischemic stroke. However, the chances to save the brain tissue by a thrombolytic therapy exponentially decrease with proceeding time after onset of symptoms.

In most cases, the beginning of the thrombolysis therapy is delayed by a variety of factors, like delivery to the hospital, re-examinations and delay of blood analysis or of CT scans. Due to this, a thrombolytic therapy is possible only in a minority of the stroke patients (2-5 %). The aim of this study is to investigate whether a "Mobile Stroke Unit", a rescue car with an integrated CT scanner, necessary for essential diagnostics, contributes to a better stroke management by saving precious time until a therapeutic decision is made. The trial is planned as a monocentric, randomised prospective trial.

DETAILED DESCRIPTION:
Stroke is the most common cause of permanent disability, the second most common cause of dementia and the third most common cause of death in elderly in industrialized countries. Approximately 85 % of all strokes are due to cerebral ischemia, whereas 15% are due to cerebral hemorrhage. In 1998, over 600.000 new strokes occurred within the European Union. Since the incidence of stroke is strongly age-related, the number of stroke victims is expected to increase substantially over the next decades as the proportion of the subjects older than 70 is estimated to grow from about 13 % to 20 % (Wahlgren 2001; The European stroke initiative, 2000). Within the next 8 years the yearly direct costs for stroke can be estimated to about 27 billion € only in Germany (Kolominsky-Rabas et al., 2006). Due to the increased incidence in the future, these costs are expected to increase by about 10 - 15 % within the next 10 years.

The main causes of ischemic stroke are thromboembolic occlusion of cerebral vessels by embolism of the heart or of the brain feeding arteries. This occlusion of a cerebral artery leads to an immediate drop of the blood flow in the corresponding arterial territory. This reduced blood flow leads to the known neurological symptoms of the affected brain area.

Animal experiments show that a massive cellular death occurs within minutes after the occlusion of an intracerebral artery in the centre of the ischemic lesion (infarction core). The region surrounding this area (penumbra) is at high risk by a functionally reduced blood flow. By improving the blood flow, this area could potentially be rescued and therefore represents the focus of every stroke therapy. Aggravatingly, the first irreversible cellular death in the penumbra starts as early as 30 minutes to 1 hour after stroke onset (Astrup et al., 1981; Heiss et al., 1983; Garcia et al., 1995; Watanabe et al., 1977; Siesjo et al., 1992; Hossmann 1994; Hu et al., 2001). Based on these data, a causal therapy of ischemic stroke appears only possible, if the cerebral blood flow is re-established within the very first hours after symptom onset (Dyker et al., 1998; Kasner et al., 1997; Adams et al., 1996; Brott et al., 1992; Del Zoppo et al., 1996; Zivin, 1998).

Currently, systemic thrombolysis with the recombinant tissue plasminogen activator (rt-PA), which is approved in Germany since 2000, represents the first evidence-based and the only causal treatment for acute ischemic stroke. The therapy should be performed as early as possible to minimize the cerebral injury and to avoid complications (i.e., hemorrhagie). Treatment with rt-PA has been studied in 6 large randomized placebo-controlled multi-centre studies (The National Institute of Neurological Disorders and Stroke rt-PA Stroke Study Group, 1995; Hacke et al. 1995; Hacke et al., 1998; Clark et al., 2000). Meta-analysis of these studies showed that a thrombolytic therapy within the first 3 hours results in a significant reduction of disability or death (Hacke et al., 1998; 2004).

The chances to save the brain tissue by a thrombolytic therapy exponentially decrease with passing time. In most cases, the patient is examined by an emergency physician, but the beginning of the final thrombolysis therapy is delayed by a variety of factors, like delivery to the hospital, neurologist re-examinations, and delay in blood analysis or CT scan.

Due to this, a therapy decision is possible within the first 3 hours only in a minority of the stroke patients. This contributes to the low lysis rate of only 4-7 % of all stroke patients.

The odds ratio (OR) of a favourable 3-month outcome of stroke therapy converges against 1 in the first 4 hours in favour of the rt-PA group (Hacke et al., 2004). Meta-analyses demonstrate that a reduction of time until the beginning of the thrombolytic therapy has the best potential to reduce the disabling effects of a stroke.

The rational of this study is to investigate whether a "Mobile Stroke Unit" contributes to a better stroke management by saving precious time until a therapeutic decision is made, according to the concept "time is brain".

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Onset of symptoms until call at least 30 min prior to the end of the approved time window for thrombolysis (and not after awakening)
* Clinical signs of ischemic stroke with suddenly occurring, measurable neurological deficits defined as impairment of language, motor function, facial palsy or asymmetry
* Patient is willing to participate voluntarily and to sign a written informed consent. Informed consent will be obtained from each patient or the subject's legally authorized representative or relative.
* Patients who are unable to sign but who are able to understand the meaning of participation in the study may give an oral witnessed informed consent. These patients have to make undoubtfully clear that they are willing to participate voluntarily and must be able to understand an explanation of the contents of the information sheet.

Exclusion Criteria:

* Age younger than 18 or older than 80 years
* Non-acute onset of symptoms
* No focal stroke-like symptoms
* Pregnant patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Time between emergency call and therapy decision

SECONDARY OUTCOMES:
Time between emergency call and end of CT, end of blood analysis, start of thrombolysis; time between symptoms and end of CT, end of blood analysis, therapy decision, number of patients with thrombolysis, start of thrombolysis, functional status

CONTACTS AND LOCATIONS:
Overall Officials: Klaus C Fassbender, Prof. Dr., Principal Investigator — Neurology, University Hospital of the Saarland, Germany
Locations (1):
- Department of Neurology, University Hospital of the Saarland, Homburg/Saar, Saarland, Germany

REFERENCES:
- [Background] Fassbender K, Walter S, Liu Y, Muehlhauser F, Ragoschke A, Kuehl S, Mielke O. "Mobile stroke unit" for hyperacute stroke treatment. Stroke. 2003 Jun;34(6):e44. doi: 10.1161/01.STR.0000075573.22885.3B. Epub 2003 May 15. No abstract available. PMID 12750527
- [Derived] Walter S, Kostopoulos P, Haass A, Keller I, Lesmeister M, Schlechtriemen T, Roth C, Papanagiotou P, Grunwald I, Schumacher H, Helwig S, Viera J, Korner H, Alexandrou M, Yilmaz U, Ziegler K, Schmidt K, Dabew R, Kubulus D, Liu Y, Volk T, Kronfeld K, Ruckes C, Bertsch T, Reith W, Fassbender K. Diagnosis and treatment of patients with stroke in a mobile stroke unit versus in hospital: a randomised controlled trial. Lancet Neurol. 2012 May;11(5):397-404. doi: 10.1016/S1474-4422(12)70057-1. Epub 2012 Apr 11. PMID 22497929